CLINICAL TRIAL: NCT06517667
Title: Efficacy and Safety of Different Hyaluronic Acid Tear Substitutes Formulations in Evaporative Dry Eye: A Randomized, Single-Blind, Comparative Study
Brief Title: Efficacy and Safety of Different Hyaluronic Acid Tear Substitutes Formulations in Evaporative Dry Eye
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, José-María Sánchez-González, Clinical professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIVIUS-ABS-003
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Patients were instructed to instill 1 drop of 0.20% Cross-linked hyaluronic acid tear substitute or 0.15% hyaluronic acid A tear substitute into each eye 3 times per day for 3 months.
Who Masked: Participant, Care Provider
Masking Description: 0.20% Cross-linked hyaluronic acid tear substitute and 0.15% hyaluronic acid tear substitute are transparent, with no special smell and the bottles were identical in appearance such that patients, investigators and care provider were masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross-linked hyaluronic acid (Experimental): Tear substitute based on 0.20% Cross-linked hyaluronic acid
  Interventions: Drug: Icross tear substitute
- Hyaluronic acid (Active Comparator): Tear substitute based on 0.15% Cross-linked hyaluronic acid
  Interventions: Drug: Hyabak tear substitute

INTERVENTIONS:
Drug: Icross tear substitute — Patients were instructed to instill 1 drop of 0.20% Cross-linked hyaluronic acid substitute into each eye 3 times per day for 3 months.
  Arms: Cross-linked hyaluronic acid
Drug: Hyabak tear substitute — Patients were instructed to instill 1 drop of 0.15% hyaluronic acid substitute into each eye 3 times per day for 3 months.
  Arms: Hyaluronic acid

SUMMARY:
The objective of the study is to compare the efficacy and safety of different hyaluronic acid tear substitutes formulations in patients with evaporative dry eye. For this purpose, a randomized, single-blind clinical trial has been designed.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported history DED.
2. Ocular surface disease index (OSDI) > 13 points.
3. Non-invasive tear film break-up time (NIBUT) < 10 s.
4. Schirmer test (ST) without anesthesia ≥ 5 mm.
5. MGD grade > 1. For MGD, the Sirius device (CSO, Florence, Italy) was used, which determines MGD grade based on loss area of meibomian glands (LAMG). MGD grade was scored from 0 to 4 (MGD grade 1 = LAMG < 25%; MGD grade 2 = LAMG ≥ 25% and < 50%; MGD grade 3 = LAMG ≥ 50% and < 75%; MGD grade 4 = LAMG ≥ 75%).

Exclusion Criteria:

1. Abnormal lid anatomy, including active blepharitis, and active lid margin.
2. All corneal disorders that affect diagnostic test, such as active corneal infection and corneal dystrophies.
3. Active ocular allergies.
4. Vectored thermal pulsation (VTP) intense pulse light (IPL), quantum molecular resonance (QMR), or other procedure to treat DED within the previous 6 months.
5. Intraocular surgery or laser ocular surgery within the previous 6 months.
6. Use of topical antibiotics and anti-inflammatory treatments, including steroids and non-steroidal anti-inflammatory drugs.
7. Systemic autoimmune diseases.
8. Contact lens wearers.
9. Pregnant or lactating women.
10. Patients who did not understand or comprehend the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Lipid layer thickness (LLT) | This outcome measure was analyzed at baseline, 1 months and 3 months.
  The Lipiview® (Johnson & JohsonVision Care, San Francisco, CA, USA) II ocular surface interferometer evaluates LLT automatically assesses LLT with nanometer precision by recording a 20 s video of the tear film interference pattern and then displays the data in interferometric color units (ICU), where1 ICU reflects approximately 1 nm of LLT.

SECONDARY OUTCOMES:
Ocular surface disease index questionnaire | This outcome measure was analyzed at baseline, 1 months and 3 months.
  The OSDI questionnaire were employed to assess the severity of DED symptoms, with scores ranging from 0 (indicating no ocular surface disease) to 100 (indicating severe ocular surface disease) points. This questionnaire was provided during consultations at each follow-up visit.
Non-invasive tear film break-up time | This outcome measure was analyzed at baseline, 1 months and 3 months.
  Tear film stability was automatically assessed using NIBUT by projecting Placido rings from the Sirius device (CSO, Florence, Italy) onto the corneal surface. The time interval between the last blink and the initial distortion of the ring pattern was defined as first NIBUT. This variable was always measured at least 12 hours after administration of the study medication and the average of 3 consecutive measurements was calculated for statistical analysis.
Schirmer I test without anesthesia | This outcome measure was analyzed at baseline, 1 months and 3 months.
  During the test, the patient is instructed to look upward while the test strip is carefully positioned between the palpebral conjunctiva of the lower eyelid and the bulbar conjunctiva. Subsequently, the patient is asked to keep their eyes gently closed for five minutes. After this period, the test strip is removed, and the Schirmer test score is determined by measuring the length of the moistened area on the strip.

CONTACTS AND LOCATIONS:
Overall Officials: José-María Sánchez-González, Study Director — University of Seville
Locations (1):
- Novovision ophthalmologic clinic, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Postorino EI, Rania L, Aragona E, Mannucci C, Alibrandi A, Calapai G, Puzzolo D, Aragona P. Efficacy of eyedrops containing cross-linked hyaluronic acid and coenzyme Q10 in treating patients with mild to moderate dry eye. Eur J Ophthalmol. 2018 Jan;28(1):25-31. doi: 10.5301/ejo.5001011. Epub 2018 Feb 19. PMID 28777385
- [Result] Posarelli C, Passani A, Del Re M, Fogli S, Toro MD, Ferreras A, Figus M. Cross-Linked Hyaluronic Acid as Tear Film Substitute. J Ocul Pharmacol Ther. 2019 Sep;35(7):381-387. doi: 10.1089/jop.2018.0151. Epub 2019 Aug 2. PMID 31373862
- [Result] Ali S, Davinelli S, Mencucci R, Fusi F, Scuderi G, Costagliola C, Scapagnini G. Crosslinked Hyaluronic Acid with Liposomes and Crocin Confers Cytoprotection in an Experimental Model of Dry Eye. Molecules. 2021 Feb 6;26(4):849. doi: 10.3390/molecules26040849. PMID 33561944
- [Result] Guarise C, Acquasaliente L, Pasut G, Pavan M, Soato M, Garofolin G, Beninatto R, Giacomel E, Sartori E, Galesso D. The role of high molecular weight hyaluronic acid in mucoadhesion on an ocular surface model. J Mech Behav Biomed Mater. 2023 Jul;143:105908. doi: 10.1016/j.jmbbm.2023.105908. Epub 2023 May 15. PMID 37209594

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT06517667/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT06517667/ICF_001.pdf